CLINICAL TRIAL: NCT00096473
Title: A 24 Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of Donepezil Hydrochloride (E2020) in Patients With Severe Alzheimer's Disease Followed by a 12 Week Open-Label Extension Period
Brief Title: Efficacy and Safety of Aricept in the Treatment of Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-315
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's Disease; dementia; acetylcholinesterase; donepezil; Aricept; memory loss; Severe dementia of the Alzheimer's type
MeSH Terms: conditions — Alzheimer Disease; Dementia; Pain; Memory Disorders | interventions — Donepezil

INTERVENTIONS:
Drug: Donepezil hydrochloride

SUMMARY:
Donepezil hydrochloride (Aricept) has been approved to treat symptoms associated with mild to moderate Alzheimer's disease (AD). Aricept has been shown to improve the memory and thinking abilities, activities of daily living and global function in patients. The purpose of the study is to further investigate the effectiveness and safety of donepezil in patients with severe Alzheimer's disease.

Donepezil is thought to work in the brain by increasing the levels of an important brain chemical called acetylcholine. This chemical helps a person's memory to work better.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed Alzheimer's Disease with MMSE score 1~12
* Have not been treated by any medication for Alzheimer's Disease in past 3 months
* Live in community or Assisted Living Facility
* Healthy or with chronic diseases that are medically controlled or stabilized
* Able to swallow tablets

Exclusion Criteria:

* Any primary neurological or psychiatric diagnosis (including depressive disorder) other than Alzheimer's Disease
* Dementia caused by organic diseases other than Alzheimer's Disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2001-01; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Assessments of global and cognitive function of Severe AD patients

SECONDARY OUTCOMES:
Assessment of behavior and performance on Activity of Daily Living in severe AD patients
Assessment of caregiver burden

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Richardson, Ph.D., Study Director — Eisai Inc.; Honglan Li, Ph.D., Study Director — Eisai Inc.
Locations (42):
- United States (28):
  - Northport, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - San Francisco, California
  - Santa Monica, California
  - Torrance, California
  - Denver, Colorado
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - North Miami, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Springfield, Massachusetts
  - Long Branch, New Jersey
  - Piscataway, New Jersey
  - New Hyde Park, New York
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Centerville, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Austin, Texas
  - Houston, Texas
- Australia (5):
  - Randwick, New South Wales
  - Brisbane, Queensland
  - Woodville South, South Australia
  - Heidelberg West, Victoria
  - Nedlands, Western Australia
- Toronto, Ontario, Canada
- Hôpital Broca-La Rochefoucauld, Paris, France
- Belfast, Ireland
- United Kingdom (6):
  - Saint Leonards-on-Sea, East Sussex
  - West End, Southampton
  - Swindon, Wilshire
  - Bath
  - Blackpool
  - Bradford